CLINICAL TRIAL: NCT05338801
Title: The Effect of Menthol on ENDS Users' Dependence, Respiratory, and Toxicants Emission Outcomes.
Brief Title: Effect of Menthol on ENDS Users' Addiction and Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA055937 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Electronic Cigarette Use
Keywords: Menthol Flavor; Tobacco Flavor
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded to study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol-flavored e-cigarette (Experimental): All participants will complete a lab visit where they will use menthol-flavored e-cigarette ad libitum for up to 60 minutes.
  Interventions: Other: Menthol-flavored e-cigarette
- Tobacco-flavored e-cigarette (Experimental): All participants will complete a lab visit where they will use tobacco-flavored e-cigarette ad libitum for up to 60 minutes.
  Interventions: Other: Tobacco-flavored e-cigarette

INTERVENTIONS:
Other: Menthol-flavored e-cigarette — All participants will complete a lab visit where they will use menthol-flavored e-cigarette ad libitum for up to 60 minutes.
  Arms: Menthol-flavored e-cigarette
Other: Tobacco-flavored e-cigarette — All participants will complete a lab visit where they will use tobacco-flavored e-cigarette ad libitum for up to 60 minutes.
  Arms: Tobacco-flavored e-cigarette

SUMMARY:
The use of electronic nicotine delivery systems (ENDS; e-cigarettes) has reached epidemic levels among young people in the United States (US). ENDS heat and vaporize a nicotine-containing liquid to produce an inhalable aerosol mist. While generally considered less harmful than combustible cigarettes, ENDS use exposes users to dependence-producing nicotine and respiratory and cardiovascular toxicants such as aldehydes. Flavor is a major factor in getting young people to use ENDS, thus limiting flavors to menthol and tobacco for prefilled cartridge ENDS "pod mods" was the first major action taken by the FDA to reduce the spread of ENDS among young people. Menthol flavor, however, can present a potential risk given its increasing popularity among young people in the US, and its puffing and nicotine-enhancing properties. Yet, the extent of menthol's ability to affect users' experience and puffing patterns, and how these affect dependence, exposure to toxicants, and clinical outcomes continue to be understudied. Such evidence will be critical to the FDA's ability to set further regulatory standards to reduce ENDS potential harm. The investigators will conduct a 2x2 (pre-post x menthol vs. tobacco flavor) crossover clinical lab study. The investigator will recruit current/past month ENDS users (n=250, 21-35 yrs), who will attend two sessions and use their ENDS once with menthol and once with tobacco flavors. The proposed studies will answer two key regulatory questions consistent with FDA's focus on the role of flavor in tobacco products' addiction and toxicity; 1) compared to tobacco flavor, does menthol carry additional risk by enhancing puffing, abuse liability, and toxicant exposure in ENDS users, and; 2) is this effect more pronounced among high dependence compared to other users. Other outcomes such as harm perception, satisfaction, clinical responses, intention to use or quit, and group comparisons such as according to race, and sex will allow the FDA a comprehensive assessment of the pros and cons of regulating mentholated ENDS for different segments of the society. Such evidence will help advance FDA regulatory policies with the potential to reduce ENDS harm.

DETAILED DESCRIPTION:
The use of electronic nicotine delivery systems (ENDS; e-cigarettes) has reached epidemic levels among young people in the US. While estimates vary, ENDS have become the leading tobacco product used by young people in this country. ENDS heat and vaporize a nicotine-containing liquid to produce an inhalable aerosol mist. While generally considered less harmful than combustible cigarettes, ENDS use exposes users to dependence-producing nicotine and other respiratory and cardiovascular toxicants such as aldehydes.

ENDS appealing design, flavors, and marketing on social media have gained them increased popularity among young people in the US. Flavor, especially, is a major driver of ENDS use among young people, thus limiting flavors for prefilled cartridge ENDS "pod mods" to menthol and tobacco was the first major action taken by the FDA to reduce the spread of ENDS. More recently, the FDA announced its commitment to banning mentholated cigarettes and cigars. Menthol ENDS, however, continue to pose a potential risk due to their increasing popularity among young people, and menthol's known initiation- and dependence-enhancing properties. Specifically, menthol can potentiate 1) inhalation by reducing irritation and allowing deeper puffs and aerosol deposition, and 2) the effect of nicotine by altering nicotinic acetylcholine receptors and increasing nicotine's bioavailability. Mentholated tobacco products, moreover, tend to affect minorities, youth, and women disproportionately. Yet, the extent of menthol's ability to alter ENDS use experience and puffing patterns, and how these affect dependence, clinical, and toxicant emissions outcomes in different users continue to be understudied.

Our team of experts in tobacco regulatory science will conduct a 2×2 (pre-post × menthol vs. tobacco flavor) crossover clinical lab study. The investigators will recruit current (past month) closed system ENDS users (n=250, 21-35 yrs, use pod-mods, or disposable ENDS), who will come to the lab for two use sessions once with menthol, and once with tobacco flavored ENDS. While the investigators apply standard lab models suitable for regulatory science, the investigators supplement them with cutting-edge puffing robot technology to explore ENDS-associated toxicant emissions (e.g., aldehydes) in the two flavor conditions. The proposed studies will answer two key regulatory-driven hypotheses consistent with this RFA's focus on the role of flavor in tobacco products' addiction and toxicity: 1) compared to tobacco flavor, does menthol carry additional risk by enhancing puffing, abuse liability, and toxicant exposure in ENDS users, and; 2) is this effect more pronounced among high dependence compared to other users. Other outcomes such as harm perception, satisfaction, respiratory symptoms and function, intention to quit or use in the future, and group comparisons according to race, and sex will provide FDA with a comprehensive assessment of the pros and cons of regulating mentholated ENDS for different users. the investigators will test these hypotheses by assessing compared to tobacco-flavored ENDS:

Aim 1. The effects of menthol flavor on subjective, puffing, and respiratory outcomes.

Aim 2. The effects of menthol flavor on ENDS toxicant emissions.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals (determined by physical examination).
* Age of 21-35 years.
* Is willing to provide informed consent.
* Is willing to attend the lab as required by the study protocol.
* E-cigarette users (defined as using e-cigarette either daily or occasionally in the past 30 days)
* Have abstained from e-cigarette use for 12 hours prior to each session

Exclusion Criteria:

* Report smoking cigarettes regularly (> 5 cigarettes/month in the past year).
* Report regular use of any other tobacco/nicotine product (e.g., e-cig, pipes, cigars) in the past year.
* Women who are breast-feeding or test positive for pregnancy (by urinalysis at screening).
* Individuals with self-reported history of chronic disease or psychiatric conditions.
* Individuals with history of or active cardiovascular disease, low or high blood pressure, seizures, and regular use of prescription medications (other than vitamins or birth control).
* Individuals that report current THC (marijuana) smoking/vaping.
* Individuals that report current EVALI or COVID-19 related symptoms (i.e., cough, shortness of breath, chest pain, nausea, vomiting, abdominal pain, diarrhea, fever, chills, or weight loss)
* Individuals that have or have been exposed to COVID-19 in the last 14 days.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Plasma nicotine | During the 2 participant visits. Blood will be taken 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Change in plasma nicotine level

SECONDARY OUTCOMES:
Minnesota Nicotine Withdrawal Scale | During participants' 2 study visits. Questionnaire will be administered 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  This scale is used to assess the extent to which product use reduces tobacco abstinence. symptoms, and consists of 11 items scored 0 - 100. These items are presented as Visual Analog Scale with item (measure) centered above a horizontal line anchored on the left with not at all and on the right with extremely.
Tiffany-Drobes Questionnaire of Smoking Urges | During participants' 2 study visits. Questionnaire will be administered 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 10 items that are scored 0 - 7. Rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Carbon monoxide levels | During participants' 2 study visits. Carbon monoxide levels will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Change in carbon monoxide levels (in parts per million).
Harm perception | During participants' 2 study visits. Questionnaire will be administered after each of the 2 e-cigarette use sessions. Each session is approximately 60 minutes ad lib use period
  This scale will assess harm perception and measure perceptions of e-cigarette. relative risk compared to cigarettes. The scale will be scored on a 7-point scale ranging from 1 (not at all harmful), to 7 (extremely harmful).
Duke Sensory Questionnaire | During participants' 2 study visits. Questionnaire will be administered after each of the 2 e-cigarette use sessions. Each session is approximately 60 minutes ad lib use period
  This scale will assess participants sensory experience of the inhaled product. The scale has nine items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
The Cigarette/ENDS Evaluation Scale (WES) | During participants' 2 study visits. Questionnaire will be administered after each of the 2 e-cigarette use sessions. Each session is approximately 60 minutes ad lib use period
  This scale assesses participants' perception of ENDS use. The scale has 11 items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
Forced expiratory volume (FEV1) | During participants' 2 study visits. FEV tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath.FEV is used to measure lung function.
Forced vital capacity (FVC) | During participants' 2 study visits. FVC tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Forced vital capacity (FVC) is the maximum amount of air that can be exhaled when blowing out as fast as possible FVC is used to measure lung function.
Peak expiratory flow (PEF) | During participants' 2 study visits. PEF tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Peak expiratory flow (PEF) is the maximal flow that can be exhaled when blowing out at a steady rate. PEF is used to measure lung function.
Forced expiratory flow | During participants' 2 study visits. Forced expiratory flow tests will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period
  Forced expiratory flow, also known as mid-expiratory flow; the rates at 25%, 50% and 75% FVC are given. Forced expiratory flowis used to measure lung function.
Puff number using eTOP topography machine | During participants' 2 study visits. Puff number is continuously measured during each e-cigarette use session (an approximately 60 minutes ad lib use period)
  Using eTOP topography machine, the investigator will assess the number of puffs during the session as part of puffing behaviour assessment.
Puff duration (seconds) using eTOP topography machine | During participants' 2 study visits. Puff duration is continuously measured during each e-cigarette use session (an approximately 60 minutes ad lib use period)
  Using eTOP topography machine, the investigator will assess the duration of the puffs (in seconds) during the session as part of puffing behaviour assessment.
Puff volume (ml) using eTOP topography machine | During participants' 2 study visits. Puff volume is continuously measured during each e-cigarette use session (an approximately 60 minutes ad lib use period)
  Using eTOP topography machine, the investigator will assess the volume of the puffs (in ml) during the session as part of puffing behaviour assessment.
Inter puff interval (IPI) (second) using eTOP topography machine | During participants' 2 study visits. Inter puff interval is continuously measured during each e-cigarette use session (an approximately 60 minutes ad lib use period)
  Using eTOP topography machine, the investigator will assess the inter puff interval (in second) during the session as part of puffing behaviour assessment.
Aldehydes (concentration) using smoking robot | During the 2 participant visits. Aldehydes will be measured 2 times in each e-cigarette use session: before and after an approximately 60 minutes ad lib use period]
  Using a smoking robot that precisely plays back the puff-by-puff behavior of each participant, we will measure concentration of aldehyde emissions during the session.

OTHER OUTCOMES:
Heart rate | During participants' 2 study visits. Heat rate will be measured from baseline continuously throughout each approximately 60 minutes session
  Change in heart rate, measured in beats per minute.
Systolic blood pressure | During participants' 2 study visits. Systolic blood pressure will be measured from baseline continuously throughout each approximately 60 minutes session
  Change in systolic blood pressure, measured in mm/hg.
Diastolic blood pressure | During participants' 2 study visits. Diastolic blood pressure will be measured from baseline continuously throughout each approximately 60 minutes session
  Change in diastolic blood pressure, measured in mm/hg.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Maziak, PhD, MD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chowdhury S, Roy S, Ferdous T, Osibogun O, Asfar T, Bursac Z, Maziak W. Menthol flavour enhances vaping experiences: a randomised crossover clinical trial. Tob Control. 2025 Aug 14:tc-2024-059202. doi: 10.1136/tc-2024-059202. Online ahead of print. PMID 40813093